CLINICAL TRIAL: NCT05573490
Title: Lifestyle Interventions for the Treatment of Early Onset Alzheimer's Disease Study
Acronym: LITES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Alzheimer's Association (Other); Tai Chi Foundation (Unknown); Alzheimer's Therapeutic Research Institute (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Dustin Hammers, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14594; AARG-22-926940 (Other Grant/Funding Number: Alzheimer's Association); 1K23AG080071-01 (NIH)
Record Dates: First submitted 2022-09-28; First posted 2022-10-10 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: lifestyle intervention; cognitive training; exercise training; cognition
MeSH Terms: conditions — Alzheimer Disease | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two conditions: (1) Computerized Cognitive Training + Tai Chi Exercise or (2) Active Control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and outcomes assessor (study coordinator) will be masked to intervention assignment. Principle investigator will not be masked given the size of the study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental Cognitive Training and Tai Chi- Qi Gong Arm (Experimental): Participants receiving 14 weeks of Cognitive Training (BrainHQ) and Tai Chi- Qi Gong exercise training
  Interventions: Device: Cognitive Training; Behavioral: Tai Chi- Qi Gong
- Active Control Arm (Active Comparator): Participants receiving 14 weeks of Brain Games (BrainHQ) and stretching
  Interventions: Device: Brain Games; Behavioral: Stretching

INTERVENTIONS:
Device: Cognitive Training — Participants will be asked to complete approximately 45 minutes of training, 4-5 sessions per week for 14 weeks (corresponding to approximately 40 hours of training total). Training will be completed via BrainHQ, a mobile application that, as used in this study, meets the FDA's definition of a medical device.
  Other Names: BrainHQ
  Arms: Experimental Cognitive Training and Tai Chi- Qi Gong Arm
Behavioral: Tai Chi- Qi Gong — Participants will be asked to complete 14 hours of training total (in 30-minute sessions, 2 days per week for 14 weeks).
  Arms: Experimental Cognitive Training and Tai Chi- Qi Gong Arm
Device: Brain Games — Participants will be asked to complete 40 hours of training total (in 45-minute sessions, 4 to 5 days per week for 14 weeks). Training will be completed via BrainHQ, a mobile application that, as used in this study, meets the FDA's definition of a medical device.
  Other Names: BrainHQ
  Arms: Active Control Arm
Behavioral: Stretching — Participants will be asked to engage in stretching exercises twice per week, for approximately 15 minutes per session. This will total of approximately 7 hours over the course of 14 weeks.
  Arms: Active Control Arm

SUMMARY:
The purpose of this study is to generate preliminary data on the benefit of computerized cognitive training and Tai Chi- Qi Gong training in participants with Early-Onset Alzheimer's Disease. It is hypothesized that participants in the experimental training condition will perform better on outcomes related to cognition, functioning, and mood at follow-up compared to participants assigned to the active control condition.

DETAILED DESCRIPTION:
This study aims to generate preliminary data regarding the efficacy of a combined cognitive-training and Tai Chi- Qi Gong exercise lifestyle intervention in participants diagnosed with Early-Onset Alzheimer's Disease (EOAD). Participants will complete a series of cognitive, functional, and mood assessments at a remotely-assessed baseline visit, and then be randomized into one of two conditions: (1) Computerized Cognitive Training + Tai Chi Exercise or (2) Active Control. Outcome measures will be repeated immediately Post-Treatment and at 6-months post-treatment Follow-Up. Specific Aim 1 will examine the feasibility of this lifestyle intervention and outcome assessments when applied to participants with EOAD. Specific Aim 2 will investigate if this lifestyle intervention improves short- and long-term cognition, functioning, and mood. Specific Aim 3 will be exploratory to assess whether individual differences in training or clinical/ demographic characteristics moderate the degree of benefit from this intervention; owing to sample size limitations in this feasibility study, focus of this latter aim will be on determining effect sizes and sample-size magnitude needed for future work.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Longitudinal Early-Onset AD Study (LEADS) parent study, and being classified via LEADS consensus criteria as having amyloid-positive Early Onset Alzheimer's Disease
* Aged 40-64 years at the time of enrollment into LEADS
* Fluent in English
* In good general health and absent another neurological disorder
* Have a knowledgeable informant.
* Have had a Clinical Dementia Rating scale of 0.5 to 1.0 at the time of enrollment into LEADS
* Have sufficient vision, hearing, comprehension, and manual dexterity to participate in the testing and training program

Exclusion Criteria:

• Have access to the internet (e.g., home, family, public library, etc.) for less than 4 hours per week

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Performance on CANTAB Connect computerized Memory Composite immediately post-intervention, after controlling for baseline performance | 15-Week Post-Intervention Follow-up
  CANTAB Connect computerized Memory Composite was selected for its remote assessment of memory, with validation in Alzheimer's Disease samples. This composite will be calculated from Paired Associates Learning, Pattern Recognition Memory, and Verbal Paired Associates subtests, with higher scores reflected better performance.
Performance on CANTAB Connect computerized Executive Composite immediately post-intervention, after controlling for baseline performance | 15-Week Post-Intervention Follow-up
  CANTAB Connect computerized Executive Composite was selected for its remote assessment of executive functioning, with validation in Alzheimer's Disease samples. This composite will be calculated from Stockings of Cambridge, Spatial Working Memory, Rapid Visual Processing, and Match To Sample subtests, with higher scores reflected better performance.
Performance on CANTAB Connect computerized Memory Composite 26 weeks after intervention, after controlling for baseline performance | 40-Week Post-Intervention Follow-up
  CANTAB Connect computerized Memory Composite was selected for its remote assessment of memory, with validation in Alzheimer's Disease samples. This composite will be calculated from Paired Associates Learning, Pattern Recognition Memory, and Verbal Paired Associates subtests, with higher scores reflected better performance.
Performance on CANTAB Connect computerized Executive Composite 26 weeks after intervention, after controlling for baseline performance | 40-Week Post-Intervention Follow-up
  CANTAB Connect computerized Executive Composite was selected for its remote assessment of executive functioning, with validation in Alzheimer's Disease samples. This composite will be calculated from Stockings of Cambridge, Spatial Working Memory, Rapid Visual Processing, and Match To Sample subtests, with higher scores reflected better performance.

SECONDARY OUTCOMES:
Benefit from Cognitive Training using Cognitive Self-Report Questionnaire immediately post-intervention, after controlling for baseline performance | 15-Week Post-Intervention Follow-up
  Cognitive Self-Report Questionnaire is a 25-item self-report questionnaire of subjective cognitive difficulties. Scores range from 0-125, with higher scores denoting greater cognitive symptoms. This measure has been used in a variety of studies examining benefit from cognitive training.
Benefit from Cognitive Training using Cognitive Self-Report Questionnaire 26 weeks after intervention, after controlling for baseline performance | 40-Week Post-Intervention Follow-up
  Cognitive Self-Report Questionnaire is a 25-item self-report questionnaire of subjective cognitive difficulties. Scores range from 0-125, with higher scores denoting greater cognitive symptoms. This measure has been used in a variety of studies examining benefit from cognitive training.
Performance on scales of functioning immediately post-intervention, after controlling for baseline performance | 15-Week Post-Intervention Follow-up
  The Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory is an informant-based rating scale that assesses the participant's ability to perform a variety of activities of daily living over the past four weeks, and has been shown to discriminate between healthy elderly controls and those with mild Alzheimer's disease. Scores range from 0-78, with higher scores denoting better functional ability.
Performance on scales of functioning 26 weeks after intervention, after controlling for baseline performance | 40-Week Post-Intervention Follow-up
  The Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory is an informant-based rating scale that assesses the participant's ability to perform a variety of activities of daily living over the past four weeks, and has been shown to discriminate between healthy elderly controls and those with mild Alzheimer's disease. Scores range from 0-78, with higher scores denoting better functional ability.
Self-reported depression immediately post-intervention, after controlling for baseline performance | 15-Week Post-Intervention Follow-up
  21-item Beck Depression Inventory-2 was used as a measure of self-reported depression. Scores range from 0-63, with higher scores denoting greater self-reported depression symptoms.
Self-reported depression 26 weeks after intervention, after controlling for baseline performance | 40-Week Post-Intervention Follow-up
  21-item Beck Depression Inventory-2 was used as a measure of self-reported depression. Scores range from 0-63, with higher scores denoting greater self-reported depression symptoms.
Self-reported quality of life immediately post-intervention, after controlling for baseline performance | 15-Week Post-Intervention Follow-up
  13-item Quality of Life- Alzheimer's Disease scale was used as a measure of self-reported quality of life. Scores range from 13-52, with higher scores denoting greater self-reported quality of life.
Self-reported quality of life 26 weeks after intervention, after controlling for baseline performance | 40-Week Post-Intervention Follow-up
  13-item Quality of Life- Alzheimer's Disease scale was used as a measure of self-reported quality of life. Scores range from 13-52, with higher scores denoting greater self-reported quality of life.
Self-reported stress immediately post-intervention, after controlling for baseline performance | 15-Week Post-Intervention Follow-up
  4-item Perceived Stress Scale was used as a measure of self-reported stress. Scores range from 0-16, with higher scores denoting greater stress.
Self-reported stress 26 weeks after intervention, after controlling for baseline performance | 40-Week Post-Intervention Follow-up
  4-item Perceived Stress Scale was used as a measure of self-reported stress. Scores range from 0-16, with higher scores denoting greater stress.
Self-reported perceived social support immediately post-intervention, after controlling for baseline performance | 15-Week Post-Intervention Follow-up
  6-Item Multidimensional Scale of Perceived Social Support (MSPSS-6) was used as a measure of self-reported support from family, friends, and a significant other. Scores range from 1-7, with higher scores denoting greater perceived social support.
Self-reported perceived social support 26 weeks after intervention, after controlling for baseline performance | 40-Week Post-Intervention Follow-up
  6-Item Multidimensional Scale of Perceived Social Support (MSPSS-6) was used as a measure of self-reported support from family, friends, and a significant other. Scores range from 1-7, with higher scores denoting greater perceived social support.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin B Hammers, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Other researchers can contact the PI to request copies of the study data.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT05573490/Prot_SAP_004.pdf
  • Informed Consent Form (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT05573490/ICF_005.pdf